CLINICAL TRIAL: NCT05597514
Title: The Application of Three-dimensional Printing High-fidelity Simulation Respiratory Models in Airway Suction and Advanced Mechanical Ventilation
Brief Title: Three-dimensional Airway Suction Model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fu Jen Catholic University (Other)
Responsible Party: Principal Investigator, Ke-Yun, Chao, Group leader of Respiratory Therapists, Fu Jen Catholic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: FJUH110116
Record Dates: First submitted 2022-10-25; First posted 2022-10-28 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-02

CONDITIONS: Satisfaction, Personal
Keywords: 3D printed; airway suction; respiratory therapy; medical education
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tranditional model group (Active Comparator): Received a regular learning
  Interventions: Other: Tranditional model education
- 3D-printed presention group (Experimental): Received a regular learning plus 3D printing model
  Interventions: Other: 3D printed educational model

INTERVENTIONS:
Other: 3D printed educational model — Slide-based presention plus 3D printed airway suction model
  Arms: 3D-printed presention group
Other: Tranditional model education — Slide-based presention plus tranditional model
  Arms: Tranditional model group

SUMMARY:
The main purpose of this study is to use 3D printing technology to high-fidelity simulation respiratory models Furthermore, the results of this study will extent to medical school and hospital.

DETAILED DESCRIPTION:
Background：

Most clinical teaching materials are expensive and inaccessible. To promote the accessibility of anatomy models and student learning effects in our medical school and hospital, we use 3D printing technology to print high-fidelity simulation respiratory models and apply them in medical education.

Study Design：

This is a single-site prospective study of medical education. Participants who are students of the School of respiratory therapy will be randomly divided into to control group and experimental group. Both groups will receive the same teaching program. The traditional education model will be used in the control group, and the 3D printed model will be used in the experimental group.

Methods：

The 3D scanning technology will be applied to create drawing files of high-fidelity simulation respiratory models, which are drawn by professional 3D drawing staff. Then, we print out the models with 3D printing technology. The output material will be close to the softness of the human models. The medical education of this study will be divided into two parts. The first part is the teaching of realistic airway suction; the second part is the simulation of advanced mechanical ventilation.

Effect：

We expect benefits that the use of 3D printing high-fidelity simulation respiratory models in medical education. For example, it can reduce the cost of education models and enhance efficacy in medical education. The experience and outcome will be shared with the medical school and hospital.

Keywords：

3D printing; medical education model; high-fidelity simulation; respiratory care.

ELIGIBILITY:
Inclusion Criteria:

* Student of Fu Jen Catholic University.

Exclusion Criteria:

* Refused to participate in the study.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2023-02-22 (Actual); Primary Completion 2023-03-08 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Examination score of pre-intervention | pre-intervention
  score of pre-intervention (maximun 100 and minimum 0), higher means a better outcome.
Examination score of post-intervention | immediately after the intervention
  score of post-intervention (maximun 100 and minimum 0), higher means a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ke-Yun Chao, PhD, Principal Investigator — Fu Jen Catholic University Hospital
Locations (1):
- Fu Jen Catholic University Hospital, Fu Jen Catholic University, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No